CLINICAL TRIAL: NCT00204035
Title: Evaluation of TEACH (Training Early Achievers for Careers in Health) Research
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13199A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Training early achievers for careers in health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Evaluation (behavior) — TEACH is a precollege enrichment program for highschool students to encourage and promote these students towards careers in clinical research. To accomplish this, instruments designed to evaluate the knowledge, attitudes, and behaviors are administered during their participation in the TEACH program.

SUMMARY:
The conceptual framework underlying the TEACH Research Program is based on a specific theoretical approach designed to influence adolescent career choice, in this case towards a career in clinical research. The factors responsible for influencing career choice that form the foundation for our investigation are: 1) the importance of role models in career choice; 2) acquisition of knowledge in order to align ambitions; and 3) the participation of students in activities that actively challenge and engage them. These three factors are addressed by the following three components of the TEACH Research Intervention: 1) participation in a research team consisting of a multi-tiered structure of mentors; 2) classroom instruction of clinical research knowledge and career strategies; and 3) a hands-on clinical research experience through an internship on the Hospitalist Project.

The evaluation of TEACH Research (Teaching Early Achievers for Careers in Health) aims to rigorously evaluate a precollege enrichment program in clinical research targeting high school students particularly underrepresented minorities, in order to increase the entry and success of these students into careers in clinical research. Through these measures, the TEACH Research Program will educate high achieving minority students and in turn hopefully encourage and promote these students to think about a career in clinical research.

DETAILED DESCRIPTION:
This projects aims to rigorously evaluate a precollege enrichment program in clinical research targeting high school students, and particularly underrepresented minorities, in order to increase the entry and success of these students into careers in clinical research.

Through the components listed in the brief summary, we hope to promote a career in clinical research among high achieving minority students. To determine whether TEACH research generates these benefits, we will recruit a larger number of candidates interested in the TEACH research than we have spots, then randomly assign students to TEACH Research or the standard more didactic enrichment programs already included in the Collegiate Scholars Program. In addition to determine the overall efficacy of the program, we will study how aspects of the program, including the didactic components, mentored research experience, and work experience, and characteristics of the student affect the development of the knowledge, attitudes, and behaviors needed for a career in clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Junior high school students in the Collegiate Scholars program

Exclusion Criteria:

* Students other than junior high school students

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: High School students
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2004-06; Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
the effect of a precollege clinical research enrichment program | 13 weeks
  We will use instruments designed to evaluate the knowledge, attitudes, and behaviors of the high school students. Written surveys will be administered test the acquisition of knowledge of clinical research and career strategies. In addition, a video assessment will be designed to elicit their attitudes towards activities designed to promote a career in clinical research, we will use peer evaluations and research team member evaluations to evaluate ability to work in teams, a key part of any research project.

SECONDARY OUTCOMES:
factors necessary for a precollege clinical research enrichment program targeting high school students to increase student interest in clinical research | 13 weeks
  We will survey students as they participate in various aspects of the program using the Experience Sampling Method (ESM). These methods will be used to survey student interest and engagement during participation in various components of the program. Also, to assess the formation of role models, we will use video-based assessments and serial evaluations of students using a tool based on the concept of a microsystem.

CONTACTS AND LOCATIONS:
Overall Officials: David Meltzer, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No